CLINICAL TRIAL: NCT01644474
Title: A Randomized, Double-Blind, Active-Controlled, Parallel-Group Study to Evaluate the Efficacy And Safety of SAR236553/REGN727 Over 24 Weeks in Patients With Hypercholesterolemia
Brief Title: Efficacy and Safety of Alirocumab (SAR236553/REGN727) Versus Ezetimibe in Patients With Hypercholesterolemia
Acronym: ODYSSEY MONO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC11716; U1111-1124-1167 (Other: UTN); 2011-001424-38 (EudraCT Number)
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ezetimibe 10 mg (Active Comparator): Oral ezetimibe 10 mg capsule daily and subcutaneous (SC) placebo injection for alirocumab every 2 weeks (Q2W) for 24 weeks.
  Interventions: Drug: Ezetimibe; Drug: Placebo (for Alirocumab)
- Alirocumab 75/Up to 150 mg Q2W (Experimental): SC injection of alirocumab 75 mg Q2W and oral placebo capsule for ezetimibe daily for 24 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
  Interventions: Drug: Alirocumab; Drug: Placebo (for Ezetimibe)

INTERVENTIONS:
Drug: Alirocumab — 1 mL subcutaneous injection in the abdomen, thigh, or outer area of the upper arm by self-injection or by another designated person using the autoinjector.
  Other Names: SAR236553; REGN727
  Arms: Alirocumab 75/Up to 150 mg Q2W
Drug: Ezetimibe — One over-encapsulated tablet orally once daily at approximately the same time of the day with or without food.
  Arms: Ezetimibe 10 mg
Drug: Placebo (for Alirocumab) — 1 mL subcutaneous injection in the abdomen, thigh, or outer area of the upper arm by self--injection or by another designated person using the autoinjector.
  Arms: Ezetimibe 10 mg
Drug: Placebo (for Ezetimibe) — One capsule orally once daily at approximately the same time of the day with or without food..
  Arms: Alirocumab 75/Up to 150 mg Q2W

SUMMARY:
Alirocumab (SAR236553/REGN727) is a fully human monoclonal antibody that binds PCSK9 (proprotein convertase subtilisin/kexin type 9).

Primary Objective of the study:

To demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) by alirocumab in comparison with ezetimibe after 24 weeks of treatment in participants with hypercholesterolemia.

Secondary Objectives:

* To evaluate the effect of alirocumab in comparison with ezetimibe on LDL-C at other time points
* To evaluate the effect of alirocumab on other lipid parameters
* To evaluate the safety and tolerability of alirocumab

DETAILED DESCRIPTION:
The maximum study duration was 34 weeks per participant, including a 24-week randomized treatment period.

ELIGIBILITY:
Inclusion criteria:

* Participants with hypercholesterolemia

Exclusion criteria:

* Age < 18 or legal age of adulthood, whichever was greater
* LDL-C < 100 mg/dL (< 2.59 mmol/L) or > 190 mg/dL (> 4.9 mmol/L)
* Fasting serum triglycerides (TG) > 400 mg/dL (> 4.52 mmol/L)
* Known history of homozygous or heterozygous familial hypercholesterolemia

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- United States (3):
  - Investigational Site Number 840603, Overland Park, Kansas
  - Investigational Site Number 840601, Cincinnati, Ohio
  - Investigational Site Number 840602, Richmond, Virginia
- Investigational Site Number 056601, Antwerp, Belgium
- Investigational Site Number 246601, Helsinki, Finland
- Netherlands (3):
  - Investigational Site Number 528602, Groningen
  - Investigational Site Number 528601, Rotterdam
  - Investigational Site Number 528603, Velp

REFERENCES:
- [Result] Roth EM, Taskinen MR, Ginsberg HN, Kastelein JJ, Colhoun HM, Robinson JG, Merlet L, Pordy R, Baccara-Dinet MT. Monotherapy with the PCSK9 inhibitor alirocumab versus ezetimibe in patients with hypercholesterolemia: results of a 24 week, double-blind, randomized Phase 3 trial. Int J Cardiol. 2014 Sep;176(1):55-61. doi: 10.1016/j.ijcard.2014.06.049. Epub 2014 Jul 2. PMID 25037695
- [Result] Roth EM, McKenney JM. ODYSSEY MONO: effect of alirocumab 75 mg subcutaneously every 2 weeks as monotherapy versus ezetimibe over 24 weeks. Future Cardiol. 2015;11(1):27-37. doi: 10.2217/fca.14.82. PMID 25606700
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 centers in 4 countries. A total of 204 participants were screened between July 2012 and November 2012, 101 of whom were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to the diabetes mellitus status. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:1 ratio ( alirocumab:ezetimibe) after confirmation of selection criteria. 103 participants were randomized.
Groups:
- Alirocumab 75/Up to 150 mg Q2W: SC injection of alirocumab 75 mg Q2W and oral placebo capsule for ezetimibe daily for 24 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when low density lipoprotein cholesterol (LDL-C) levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
Period: Overall Study
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Started | 51 (Randomized) | 52 (Randomized)
Treated | 51 | 52
Completed | 44 | 44
Not Completed | 7 | 8
Not completed — Poor compliance to protocol | 1 | 0
Not completed — Consent withdrawn by participant | 0 | 1
Not completed — Participant moved | 0 | 1
Not completed — Adverse Event | 4 | 5
Not completed — Site scheduling error | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ezetimibe 10 mg: Oral ezetimibe 10 mg capsule daily and SC placebo injection for alirocumab Q2W for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (5.3) | 60.8 (4.6) | 60.2 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 27 | 28 | 55
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Calculated LDL-C in mmol/L from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/2.2]).
  mmol/L | 3.58 (0.6) | 3.65 (0.7) | 3.62 (0.7)
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C in mg/dL from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/5]).
  mg/dL | 138.3 (24.5) | 141.1 (27.1) | 139.7 (25.8)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-Treat (ITT) Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -15.6 (3.1) | -47.2 (3.0)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; Alirocumab group was compared to ezetimibe group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -31.6, 95% CI 2-sided [-40.2 to -23.0] — Alirocumab vs Ezetimibe

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -19.6 (2.6) | -48.1 (2.6)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -28.5, 95% CI 2-sided [-35.7 to -21.2] — Alirocumab vs Ezetimibe

3. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 46 | 48
percent change | -11.0 (2.4) | -36.7 (2.3)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -25.8, 95% CI 2-sided [-32.3 to -19.2] — Alirocumab vs Ezetimibe

4. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -15.1 (2.9) | -40.6 (2.8)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -25.5, 95% CI 2-sided [-33.5 to -17.4] — Alirocumab vs Ezetimibe

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -10.9 (2.2) | -29.6 (2.1)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -18.7, 95% CI 2-sided [-24.7 to -12.7] — Alirocumab vs Ezetimibe

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Apo-B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 46 | 48
percent change | -11.7 (2.1) | -37.3 (2.1)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -25.7, 95% CI 2-sided [-31.5 to -19.8] — Alirocumab vs Ezetimibe

7. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 24
Population: non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -16.7 (2.4) | -42.5 (2.3)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -25.8, 95% CI 2-sided [-32.4 to -19.2] — Alirocumab vs Ezetimibe

8. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 24
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -12.0 (1.7) | -30.3 (1.7)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -18.3, 95% CI 2-sided [-23.1 to -13.5] — Alirocumab vs Ezetimibe

9. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percentage of participants | 32.2 | 88.1
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 34.8, 95% CI 2-sided [8.7 to 139.0] — Alirocumab vs Ezetimibe

10. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percentage of participants | 2.4 | 59.4
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0001, Regression, Logistic — Threshold for significance was ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 69.8, 95% CI 2-sided [8.8 to 556.0] — Alirocumab vs Ezetimibe

11. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from a multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -12.3 (3.8) | -16.7 (3.7)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Alirocumab 75/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4013, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -4.4, 95% CI 2-sided [-14.8 to 5.9] — Alirocumab vs Ezetimibe

12. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | 1.6 (1.9) | 6.0 (1.9)

13. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 24
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | 1.6 (2.0) | 9.0 (2.0)

14. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -14.2 (3.7) | -17.2 (3.7)

15. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -10.8 (4.3) | -11.9 (4.2)

16. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: as for outcome 14
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 51 | 52
percent change | -2.3 (3.5) | -12.2 (3.4)

17. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-1) at Week 24 - ITT Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment (Apo A-1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 46 | 48
percent change | -0.6 (1.6) | 4.7 (1.6)

18. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 24
Population: Apo A-1 ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up to 150 mg Q2W
Number analyzed (Participants) | 46 | 48
percent change | -2.2 (1.4) | 2.3 (1.4)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 32 post-treatment follow-up visit) regardless of seriousness or relationship to study drug.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment-emergent period' (from the first dose of double-blind study drug administration (capsule or injection, whichever came first) up to the day of the last double-blind injection + 70 days).
Groups:
- Ezetimibe 10 mg: Participants exposed to Ezetimibe 10 mg (mean exposure of 22 weeks).
- Alirocumab 75/Up150 mg Q2W: Participants exposed to Alirocumab 75 mg/Up to 150 mg Q2W (mean exposure of 22 weeks).
Arm/Group | Ezetimibe 10 mg | Alirocumab 75/Up150 mg Q2W
Serious Adverse Events (participants affected / at risk) | 1/51 | 1/52
Other Adverse Events (participants affected / at risk) | 27/51 | 25/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ezetimibe 10 mg (N=51) | Alirocumab 75/Up150 mg Q2W (N=52)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ezetimibe 10 mg (N=51) | Alirocumab 75/Up150 mg Q2W (N=52)
Nasopharyngitis (Infections and infestations) | 8 | 12
Influenza (Infections and infestations) | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Urinary tract infection (Infections and infestations) | 3 | 0
Headache (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
Due to administrative error in the automated process (which was detected after database lock), planned dose up-titration criteria for LDL-C levels was changed from ≥100 mg/dL to ≥70 mg/dL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.